CLINICAL TRIAL: NCT02697331
Title: Evaluation of the Role of Vaginal Progesterone in Prevention of Preterm Labor in Twin Gestation With Short Cervix: Randomised Controlled Trial
Brief Title: Vaginal Progesterone in Twin With Short Cervix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Reda, DR, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AIN-2222-RCT
Record Dates: First submitted 2016-02-27; First posted 2016-03-03 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Preterm Birth; Twin Dichorionic Diamniotic Placenta
Keywords: Short cervix, twins, progesterone
MeSH Terms: conditions — Premature Birth | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- progesterone (Active Comparator): 74 patients will receive progesterone pessary 200mg twice daily
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator): 74 patients will receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Progesterone — women will receive progesterone vaginal pesarries containing 200mg of progesterone twice daily . it will be used by the patient as one vaginal pessary per vagina twice per day .
  women will be showed how to use tablets . medication will be started at 20 -24 weeks and stopped at 36+6 weeks
  Other Names: uterocare
  Arms: progesterone
Other: Placebo — women will receive placebo pessary twice a day. women will be showed how to use tablets . medication will be started at 20-24 weeks and stopped at 36+6 weeks
  Arms: Placebo

SUMMARY:
Aim of the work The aim of this study is to assess the efficacy of the use of vaginal progesterone as a method of prevention of preterm labour in twin gestations with short cervix .

Study Design:

The study is designed as randomized ,placebo-controlled, clinical trial . All women with dichorionic diamniotic twin pregnancy will be followed up in the antenatal care at the out patient clinic. Randomization of cases will be done by computer method . 156 women with dichorionic diamniotic twin pregnancy and cervical length 10mm to 25mm detected on transvaginal sonogram between 20w to 24w gestational age were enrolled in the study and were distributed in two groups:group P (cases ) and group N (controls) . The randomization allocation was 1 : 1 (vaginal progesterone capsule : placebo).

DETAILED DESCRIPTION:
Aim of the work The aim of this study is to assess the efficacy of the use of vaginal progesterone as a method of prevention of preterm labour in twin gestations with short cervix .

Study Design:

The study is designed as randomized ,placebo-controlled, clinical trial . All women with dichorionic diamniotic twin pregnancy will be followed up in the antenatal care at the out patient clinic. Randomization of cases will be done by computer method . 156 women with dichorionic diamniotic twin pregnancy and cervical length 10mm to 25mm detected on transvaginal sonogram between 20w to 24w gestational age were enrolled in the study and were distributed in two groups:group P (cases ) and group N (controls) . The randomization allocation was 1 : 1 (vaginal progesterone capsule : placebo).

Inclusion Criteria :

( All pregnant women known to have Dichorionic Diamniotic twins diagnosed on 12 week dating scan will be offered transvaginal ultrasound scan to assess cervical length at 20-24 week anomaly scan ) and so inclusion criteria include:

1. ( Dichorionic Diamniotic twins ) and both twins are living .
2. (Short Cervix 10-25mm) Diagnosed by transvaginal ultrasound scan between 20-24 weeks

Exclusion Criteria :

1. Cervical cerclage in place or planned .
2. on tocolytic drugs .
3. medically indicated preterm delivery < 35w of gestation .
4. known allergy to progesterone or peanuts ( as the active treatment contain peanut oil) .
5. known contraindication to progesterone

   1. Liver dysfunction or disease
   2. Known or suspected malignancy of breast or genital organs
   3. Active thromboembolic disorder , or history of hormone-associated thromboembolic disorder
6. known major structural or chromosomal fetal abnormality .
7. Rupture of fetal membranes (leakage of amniotic fluid one or both sacs).

ELIGIBILITY:
Inclusion Criteria:

* ( All pregnant women known to have Dichorionic Diamniotic twins diagnosed on 12 week dating scan will be offered transvaginal ultrasound scan to assess cervical length at 20-24 week anomaly scan ) and so inclusion criteria include:

  1. ( Dichorionic Diamniotic twins ) and both twins are living .
  2. (Short Cervix 10-25mm) Diagnosed by transvaginal ultrasound scan between 20-24 weeks .

Exclusion Criteria:

1 - Cervical cerclage in place or planned . 2- on tocolytic drugs . 3- medically indicated preterm delivery < 35w of gestation . 4- known allergy to progesterone or peanuts ( as the active treatment contain peanut oil) .

5- known contraindication to progesterone

1. Liver dysfunction or disease
2. Known or suspected malignancy of breast or genital organs
3. Active thromboembolic disorder , or history of hormone-associated thromboembolic disorder 6- known major structural or chromosomal fetal abnormality . 7- Rupture of fetal membranes (leakage of amniotic fluid one or both sacs)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
delivery at <37weeks of gestation | 37 weeks gestation determined by 12 weeks dating scan
  Preterm birth

SECONDARY OUTCOMES:
adverse neonatal outcome | From date of delivery to date of hospital discharge up to 28 days
  admission/Hypoglycaemia/Respiratory distress/feeding difficulty/sepsis
preterm Delivery for different gestational age | less than 28 weeks, 28- 32 weeks, 32-34weeks, 34-37 weeks
  preterm delivery
Maternal adverse effects | From randomization at 20-24 weeks till 37 weeks or delivery whichever occurs sooner
  Drug adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelhafeez, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Maternity Hospital, Cairo, Egypt